CLINICAL TRIAL: NCT04627727
Title: Effect of a Low FODMAP Diet on SIBO Breath Test Positivity
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Early termination due to lack of funds, staffing
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Judy Nee, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000622
Record Dates: First submitted 2020-10-30; First posted 2020-11-13 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: SIBO
MeSH Terms: interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low FODMAP diet (Experimental): Consenting patients fulfilling the inclusion and exclusion criteria will undergo a 7-day screening period to assess baseline symptoms and then go on a 4-week low FODMAP diet
  Interventions: Other: low FODMAP diet

INTERVENTIONS:
Other: low FODMAP diet — low FODMAP diet

SUMMARY:
Bloating is the most common symptom associated with disorders of brain-gut interaction (i.e., functional bowel disorders) such as irritable bowel syndrome, a disorder characterized by abdominal pain and altered bowel habits which affects up to 11% of world population. A common cause of bloating is small intestinal bacterial overgrowth (SIBO), a condition defined by excessive and/or abnormal type of bacteria in the small bowel. The potential role of SIBO for irritable bowel syndrome (IBS) was initially proposed by Pimentel et al. Using lactulose breath tests (LBTs), 78% of patients with IBS were also diagnosed with SIBO. After antibiotic therapy, 48% of patients no longer met the Rome criteria for IBS. A recent systematic review and meta-analysis concluded that the prevalence of SIBO is increased in IBS.

DETAILED DESCRIPTION:
Despite the clinical efficacy of LFD in improving symptoms of IBS-D, its mechanism of action is not clear. Recently, Zhou et al have shown FODMAPs induce colonic tight junction dysfunction and visceral hypersensitivity in rat models, both of which are reversible when rats were fed an LFD. They further showed that this effect of FODMAPs is mediated by microbial dysbiosis and elevated fecal lipopolysaccharide level. However, studies evaluating the effect of LFD on colonic permeability of humans are lacking. Studies have shown significant differences in intra-individual luminal and mucosal microbiome of patients with functional gastrointestinal disorders as well as an increase in Prevotella abundance in IBS patients with SIBO as compared with IBS patients without SIBO. Thus, the exact effect of FODMAP on intestinal permeability and mucosal microbiome in humans is not clear and needs further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years at the time of screening
* Meet Rome IV criteria for functional bloating
* IBS-SSS score of at 176 (0-500)
* SIBO positive

Exclusion Criteria:

* individuals already on a LFD or other dietary restriction such as gluten free diet within the past 6 months
* individuals with peanut, soy, or seafood allergies or insulin-dependent diabetes
* known history of celiac disease, inflammatory bowel disease or microscopic colitis
* prior small bowel or colonic surgery or cholecystectomy
* pregnant patients
* antibiotics, excluding topical, in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Lembo, M.D, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemos MPC, Zucoloto TG, Oliveira MC, de Oliveira GLV. Dysbiosis and Gut Microbiota Modulation in Systemic Sclerosis. J Clin Rheumatol. 2022 Mar 1;28(2):e568-e573. doi: 10.1097/RHU.0000000000001748. PMID 34030162

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low FODMAP Diet
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: SIBO positive participants who undergo 3 weeks of low FODMAP diet
Groups:
- SIBO Positive Patients: SIBO positive patients who undergo 3 weeks of Low FODMAP diet
Arm/Group | SIBO Positive Patients
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants] — age determined by date of birth
  Participants
    <=18 years | 0
    Between 18 and 65 years | 14
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  white, non-hispanic | 12
  asian | 2
SIBO positive [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: SIBO Diagnosis
Description: Number of Participants with Negative and Positive SIBO
Time Frame: four weeks
Population: Participants with SIBO positivity, then underwent 4 weeks of LOW FODMAP diet and repeated SIBO breath test at end of study.
Measure: Number; unit: participants
Arm/Group | Low FODMAP Diet
Number analyzed (Participants) | 14
participants
  Participants with negative SIBO Diagnosis | 10
  Participants with Positive SIBO Diagnosis | 4

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Low FODMAP: low FODMAP x 3 weeks
Arm/Group | Low FODMAP
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT04627727/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04627727/ICF_001.pdf